CLINICAL TRIAL: NCT00371670
Title: A Phase II, 12-month, Double-blind, Placebo-controlled, Dose-finding, Multicenter Study to Evaluate the Safety, Tolerability, and Disease Modifying Efficacy of Daily Oral AAE581 (10, 25 and 50 mg Tablets) in Patients With Painful Knee Osteoarthritis, Kellgren-Lawrence Grade 3 by X-ray
Brief Title: Safety/Efficacy of Balicatib (AAE581) in Adults With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE581C2201
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Knee Osteoarthritis
Keywords: Knee, osteoarthritis, pain, disease modifying
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — balicatib

INTERVENTIONS:
Drug: balicatib (AAE581)

SUMMARY:
This study will test efficacy and safety of AAE581 compared to placebo in limiting cartilage loss in patients with painful knee osteoarthritis which is confirmed by X-ray

ELIGIBILITY:
Inclusion Criteria:

* At least one knee with osteoarthritis with Kellgren-Lawrence grade 3
* Significant osteoarthritis pain in the knee
* Presence of at least one of the risk factors: obesity (BMI > 28), osteoarthritis at other sites, knee effusion, family history of total joint replacement

Exclusion Criteria:

* Women with childbearing potential
* Secondary osteoarthritis
* Treatment with intra-articular or systemic steroids
* Inability to undergo MRI acquisition

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2004-12; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in knee cartilage volume in the target compartment after 6 months

SECONDARY OUTCOMES:
Change from baseline in:
- Cartilage volume in the different regions of the knee after 6 and 12 months,
- Cartilage score (Whole Organ MRI Scoring system (WORMS)) in the different regions of the knee after 6 and 12 months,
- Bone marrow edema score (WORMS) in the different regions of the knee after 6 and 12 months,
- Joint space width after 6 and 12 months,
- Markers of bone and cartilage degradation (CTX-I and CTX-II at 3, 6, 9, and 12 months
- Pain (analgesic consumption, Western Ontario and McMaster Universities Osteoarthritis Index, Visual Analogue Scale, criteria of the Outcome Measures in Rheumatology Osteoarthritis-Research Society International at 1, 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Pinnacle Research Group, Anniston, Alabama, United States
- Novartis, Nuremberg, Germany